CLINICAL TRIAL: NCT05637242
Title: Ventricular Assist Device (VAD) Research Registry and Blood Sub-Study
Status: Terminated | Type: Observational
Why Stopped: Study was not able to achieve primary objective and there is no intention to work towards its achievement
Sponsor: Corewell Health West (Other)
Responsible Party: Principal Investigator, Renzo Loyaga Rendon, Renzo Loyaga Rendon MD, Corewell Health West
Other Study IDs: 2015-073
Record Dates: First submitted 2016-04-19; First posted 2022-12-05 (Actual); Last update posted 2024-06-05 (Actual); Status verified 2024-06

CONDITIONS: Heart Failure
Keywords: Ventricular Assist Device
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — Biospecimen retained include blood and serum.
Oversight: Data Monitoring Committee: No

SUMMARY:
This study is meant to predict the outcome of VAD therapy, by forming a VAD registry for quality assessment, research, and real-time monitoring of patients on VAD therapy. The goal is to optimize the use of VAD therapy for patients, to create an online quality measurement tool for VAD treatment, and to create algorithms to estimate the prognosis for patients getting a VAD.

DETAILED DESCRIPTION:
Patients eligible for VAD are being sampled before surgery for plasma as well as peripheral blood cells. After surgery patients are being sampled again at 24 h and 7 days. Inflammatory response is being monitored on gene expression as well as cell level and on cytokine level in relation to the outcome.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is ≥ 18 years of age
2. Subject is treated with a VAD at the Butterworth Campus, Spectrum Health.

Exclusion Criteria:

1. Subject is less than 18 years of age.
2. Known prisoners of the state.
3. Subject is pregnant.
4. Non- English speaking patients will be excluded from the blood sub-study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients being implanted with a ventricular assist device.
Sampling Method: Non-Probability Sample
Enrollment: 371 (Actual)
Dates: Start 2016-02; Primary Completion 2021-10-13 (Actual); Study Completion 2024-05-29 (Actual)

PRIMARY OUTCOMES:
One year mortality | One year
  Mortality will be assessed yearly.

SECONDARY OUTCOMES:
Cytokine Analysis | Pre-implant, within 24 hours of implant, and 7 days post-implant
Inflammatory cell subtype | Pre-implant, within 24 hours of implant, and 7 days post-implant
Hospital readmissions | Will be assessed yearly until death or explant

CONTACTS AND LOCATIONS:
Overall Officials: Renzo Loyaga, MD PhD, Principal Investigator — The DeVos Cardiovascular Research Program, Frederik Meijer Heart & Vascular Institute, Corewell Health
Locations (1):
- Frederik Meijer Heart Center, Grand Rapids, Michigan, United States

IPD SHARING:
Plan to Share IPD: No